CLINICAL TRIAL: NCT01478919
Title: Risk Factors for Local Residual Neoplasia After Convetional Endoscopic Mucosal Resection of Laterally Spreading Tumors
Brief Title: Risk Factors for Residual Neoplasia After Endoscopic Mucosal Resection
Status: Completed | Type: Observational
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Premysl Falt MD, Investigator, Vitkovice Hospital
Other Study IDs: DDC VN 02
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
Keywords: Endoscopic Mucosal Resection; Laterally Spreading Tumor; Local Residual Neoplasia; Colonoscopy; Therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Laterally Spreading Tumors (LST) are important precursosrs of invasive colorectal cancer. Endoscopic treatment has replaced surgery in most of the cases. Nevertheless, after conventional Endoscopic Mucosal Resection (CER), Local Residual Neoplasia (LRN) is an issue. Therefore, endoscopic follow-up and treatment are necessary. To decrease its occurrence, the risk factors of LRN shoudl be identified. Thereafter, in high-risk patients, other modalities of initial treatment including Endoscopic Submucosal Dissection (ESD) and surgical treatment, could be considered. The purpose of this prospective study is to identify risk factors associated with the presence of LRN after CER of LSTs.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients referred for EMR of LST

Exclusion Criteria:

* polyposis syndromes
* previous therapeutic attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for Endoscopic Mucosal Resection (EMR) of Laterally Spreading Tumors (LST.)
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Occurence of Local Residual Neoplasia (LRN) | 3 months
  LRN was defined as a histologically confirmed neoplastic tissue in the biopsy samples obtained from post-resection scar during follow-up colonoscopy 3 months after endoscopic resection

SECONDARY OUTCOMES:
Evaluation of Selected Risk Factors for Local Residual Neoplasia (LRN) | 3 months
  Evaluation of selected patient- and lesion-related risk factors associated with LRN (gender, age, lesion size, location, morphology, pit pattern, histology, type of resection, and others)

CONTACTS AND LOCATIONS:
Locations (1):
- Vitkovice Hospital, Ostrava, Czechia

REFERENCES:
- [Background] Urban O, Kijonkova B, Kajzrlikova IM, Vitek P, Kliment M, Fojtik P, Falt P, Reiterova K, Horava V Jr. Local residual neoplasia after endoscopic treatment of laterally spreading tumors during 15 months of follow-up. Eur J Gastroenterol Hepatol. 2013 Jun;25(6):733-8. doi: 10.1097/MEG.0b013e32835eda96. PMID 23442418